CLINICAL TRIAL: NCT05063760
Title: Exercise in Prevention & Treatment of Chemotherapy-related Late Toxicity in Testicular Germ Cell Cancer Survivors: the Role of Skeletal Muscle
Brief Title: Exercise in Testicular Germ Cell Cancer Survivors
Acronym: ExCell
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Slovak Academy of Sciences (Other Government)
Collaborators: Comenius University (Other)
Responsible Party: Principal Investigator, Jozef Ukropec, PhD, DSc, Slovak Academy of Sciences
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2/0164/20; SRDA19-0411 (Other Grant/Funding Number: Slovak Research and Development Agency)
Record Dates: First submitted 2021-03-18; First posted 2021-10-01 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-12

CONDITIONS: Testicular Germ Cell Tumor
Keywords: TGCT; exercise intervention; Magnetic resonance spectroscopy; skeletal muscle; chemotherapy-induced metabolic toxicity
MeSH Terms: conditions — Testicular Germ Cell Tumor

STUDY DESIGN:
Intervention Model Description: controled trial with exercise intervention
Who Masked: Investigator, Outcomes Assessor
Masking Description: lab technicians and statistician are blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TGCT patients - exercise (Experimental): TGCT survivors, men, 25-55 yrs old, 3 and more years after successful treatment of TGCT, with the capacity to undergo aerobic-strength intervention assessed by cardiologist
  Interventions: Behavioral: aerobic-strength exercise intervention (6-months)
- TGCT patients - nonexercising controls (No Intervention): TGCT survivors, men, 25-55 yrs old, 3 and more years after successful treatment of TGCT, with the capacity to undergo aerobic-strength intervention assessed by cardiologist

INTERVENTIONS:
Behavioral: aerobic-strength exercise intervention (6-months) — 6 month supervised exercise intervention in TGCT survivors (1 hour sessions 3 x per week),
  Arms: TGCT patients - exercise

SUMMARY:
Regular exercise is effective in prevention & treatment of chronic diseases. Exercise can reduce late toxicity of chemotherapy, commonly found in cancer survivors, which is yet to be translated into clinical practice.

Mechanisms of exercise benefits in oncologic patients are far from being elucidated, and include increase in muscle mass, reduction of fat mass, systemic inflammation and cardiometabolic risk. Synchronization of exercise adaptive response is, to an extent, mediated by bioactive molecules released from muscle, with anti-inflammatory & tumor-suppressing properties. Muscle satellite cells are a source of regeneration, muscle structural integrity & functional capacity. Phenotypes of muscle cells, such as secretory profile, lipid & glucose metabolism, mirror clinical phenotypes of the donor. Importantly, muscle cells' metabolism in vitro can be modulated by 8-12 week training in vivo. Epigenetic mechanisms regulating muscle & systemic metabolism in cancer survivors are not yet understood.

DETAILED DESCRIPTION:
Aims:

* To assess the impact of 6-month supervised, individualized aerobic-strength exercise training intervention in cancer survivors with chemotherapy-induced late toxicity . (i) on the whole-body energy and glucose metabolism, anthropometric parameters, physical fitness & activity profile, motor functions and quality of life in testicular germ cell cancer (TGCC) survivors, more than 3 years after cisplatin-based chemotherapy; with the 2-year follow up; . (ii) on skeletal muscle mass, morphology as well as functional and metabolic state detected in vivo (31P-MR spectroscopy).

(iii) on metabolic characteristics of primary skeletal muscle cells;

* To determine the impact of exercise intervention on circulating bioactive molecules (exerkines), putative mediators of exercise health benefits as well as on levels of circulating inflammatory cytokines, which likely contribute to the pathogenesis of chemotherapy-induced late toxicity;
* To evaluate the role of (a) selected exercise-regulated bioactive molecules, (b) exercise-mimicking treatment (by electric pulse stimulation) and (c) cisplatin treatment on metabolism and mitochondrial function of differentiated human muscle cells in culture;
* To investigate the associations between intervention-induced shifts in circulating bioactive molecules and selected metabolic, anthropometric and motor parameters.

The generated results will enable us (i) to gain a better insight into pathomechanisms of muscle-associated chemotherapy-induced late toxicity and the role of skeletal muscle & systemic mediators in the exercise-induced health benefits in TGCC survivors; and (ii) to validate the effectiveness of the individually-tailored exercise intervention in reducing chemotherapy-related toxicity in patients with TGCC, with the aim to transfer this knowledge into clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* TGCT survivors, with chemotherapy-induced metabolic toxicity, men, 25-55 years old, with the capacity to undergo training, signed written informed consent

Exclusion Criteria:

* serious / uncontrolled chronic diseases, non-compliance, other health issues as assessed by oncologists / investigators

Ages: 25 Years to 55 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-01-15 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
change in the glucose tolerance | parameter will be measured before and after 6 month intervention
  change in glucose tolerance (as measured by oral glucose tolerance test)
change in resting energy expenditiure and metabolic substrate preference | parameters will be measured twice before and after 6 month intervention
  change in resting energy expenditure calculated by Weir equation from VO2 and metabolic substrate preference RQ VCO2/VO2 (as measured by indirect calorimetry)
change anthropometric parameters of obesity | parameters will be measured twice before and after 6 month intervention
  BMI (kg.m-2) , fat mass (% electric bioimpedance), lean body mass (% electric bioimpedance), visceral adiposity (%, elecgtric bioimpedance)
change physical fitness | parameter will be measured twice before and after 6 month intervention
  VO2max (mlO2 per kg BW min) as measured by bicycle spiroergometry

SECONDARY OUTCOMES:
change in quality of life for cancer patients | measured twice before and after 6 month intervention
  validated questionnaire
change in muscle strength | measured twice before and after 6 month intervention
  dynamometry
change in cognitive functions | measured twice before and after 6 month intervention
  standardised cognitive test Cogstate

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Ukropcova, MD, PhD, Prof, Principal Investigator — Biomedical Research Center, Slovak Acad Sci
Locations (2):
- Slovakia (2):
  - National Cancer Institute, Bratislava, Please Select
  - Biomedical Research Center Slovak Academy of Sciences, Bratislava, Please Select

IPD SHARING:
Plan to Share IPD: No
we will share IPD upon reasonable request